CLINICAL TRIAL: NCT04019054
Title: Transcranial Magnetic Stimulation (TMS) in Conjunction With Exposure Therapy for the Treatment of Spider Phobia
Brief Title: TMS and Exposure Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael K Leuchter, Medical Student, David Geffen School of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-000218
Record Dates: First submitted 2019-07-07; First posted 2019-07-15 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Arachnophobia; Phobia
Keywords: Transcranial Magnetic Stimulation (TMS); Exposure Therapy; Phobia; Intermittent Theta-Burst Stimulation (iTBS)
MeSH Terms: conditions — Arachnophobia; Phobic Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the study treatment (iTBS stimulation to the ventromedial prefrontal cortex) or control treatment (iTBS stimulation to the vertex). Treatments will occur immediately following exposure therapy (both groups will undergo identical exposure therapy), and groups will receive iTBS to the same site for all three treatments
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assignment will be performed randomly and tracked by clinical staff involved with the TMS treatment itself, and research staff assessing outcomes and analyzing data will be blinded to groups until after analysis is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) (Experimental): Stimulation intensity of 100% of the individual resting motor threshold in bursts of three pulses at a frequency of 50 Hz every 200 ms on top of a 5Hz carrier wave. Pulse delivery is over 2 s and repeated every 10 s, 20 times in succession, for a total of 600 pulses delivered in 3.33 minutes.
  Delivered over vmPFC, as determined by position Fpz of the international 10-20 EEG electrode system.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS), Ventromedial Prefrontal Cortex (vmPFC)
- Control iTBS, vertex (Placebo Comparator): Stimulation intensity of 100% of the individual resting motor threshold in bursts of three pulses at a frequency of 50 Hz every 200 ms on top of a 5Hz carrier wave. Pulse delivery is over 2 s and repeated every 10 s, 20 times in succession, for a total of 600 pulses delivered in 3.33 minutes.
  Delivered over vertex, as determined by position Cz of the international 10-20 EEG electrode system.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS), vertex

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation (iTBS), Ventromedial Prefrontal Cortex (vmPFC) — iTBS delivered to vmPFC for active treatment of spider phobia.
  Arms: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC)
Device: Intermittent Theta Burst Stimulation (iTBS), vertex — iTBS delivered to vertex for placebo treatment of spider phobia.
  Arms: Control iTBS, vertex

SUMMARY:
Spider phobia is an exceedingly common phobia throughout the world. The current standard treatment involves exposure therapy, which consists of a series of brief exposures of an individual to the thing they fear, in this case spiders. This study aims to examine the use of a neuromodulatory technology, transcranial magnetic stimulation (TMS), as a possible treatment option for spider phobia. TMS uses low-intensity electromagnetic energy to stimulate the brain, introducing energy into critical hubs of brain networks to "reset" their function and alleviate symptoms with very few side-effects.

This study will consist of four separate visits. After screening subjects for spider phobia, baseline testing of subjective distress measures and physiologic stress data (heart rate variability and sweat response) during a prolonged spider exposure test will be collected. Subjects will then be placed into one of two groups: one receiving exposure therapy and intermittent Theta Burst Stimulation (iTBS) TMS (active study group), and another receiving exposure therapy with iTBS to a circuit not involved in a phobic reaction (control study group). Subjects will undergo their first treatment session during the first visit following the baseline data collection; the second and third treatments will occur the following two days. The fourth visit will occur one week after the third and consist of the same testing as the first visit; the same data will be collected. Changes from pre- to post-treatment in both subjective and physiologic data will be compared between the treatment and sham groups to examine effects of TMS on spider phobia.

DETAILED DESCRIPTION:
OVERVIEW The experiment will consist of four days. Day 1 will include informed consent, questionnaires, a behavioral approach test with a spider, a series of short exposures with a spider, and the first TMS treatment (for a total of approximately 75-90 minutes). Day 2 will occur one to two days after Day 1 and will consist of a second series of short exposures with a spider and the second TMS treatment (30 minutes). Day 3 will occur one to two days after Day 2 and will also consist of a series of short exposures and a TMS treatment (30 minutes). Day 4 will occur five to seven days after Day 3 and will consist of post-study questionnaires and an identical behavioral approach test as is conducted on the first visit (30 minutes). Participants will be randomized to either an active TMS treatment group (using an iTBS stimulation protocol over the participant's ventro-medial prefrontal cortex, an area involved in phobic response) or a control TMS treatment group (using the same iTBS stimulation protocol over the central sulcus and between hemispheres, a site not associated with memory or fear response).

Prospective participants will be recruited from two groups: 1) undergraduate students recruited through the UCLA Psychology Department Subject Pool (i.e., SONA) and 2) general population over the age of 18 recruited via flyers. All prospective participants will be screened with the 31-question Spider Phobia Questionnaire (SPQ) to ensure eligibility for participation, with a minimum total score equal to or greater than 17 required for participation.(Klorman, Weerts, Hastings, Melamed, & Lang, 1974) Participants will be enrolled for the study only if they are able to complete all four visits of the experiment. Exclusion criteria will include:

1. Subject is mentally or legally incapacitated, unable to give informed consent.
2. Subjects with psychosis (psychotic depression, schizophrenia, or schizoaffective diagnoses (lifetime)); bipolar disorder (lifetime); dementia (lifetime); delirium within the past 6 months; eating disorder within the past year; obsessive-compulsive disorder (lifetime); post-traumatic stress disorder within the past year; acute risk for suicide or self-injurious behavior. Patients with diagnostic uncertainty or ambiguity (e.g. rule-out pseudodementia of depression) will be excluded.
3. Subjects with a HamD suicidality item score of '3' or '4,' corresponding to "suicidal ideas or gestures" or "attempts at suicide," will be excluded.
4. Subjects with exposure to ECT within the past 6 months, previous TMS treatment for any condition, or VNS treatment (lifetime).
5. Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke, CVA, or TIAs; cerebral aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.
6. Any history of intracranial implant including cochlear implant, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments; implanted cardiac pacemaker, defibrillator, vagus nerve stimulator, deep brain stimulator; or other implanted devices or objects contraindicated by product labeling.
7. Neurological conditions including epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, history of repetitive or severe head trauma, or with primary or secondary tumors in the CNS.
8. current pregnancy or breast feeding.
9. Infection or loss of integrity of skin over the forehead, where the device will be positioned.
10. Increased risk of seizure as indicated by: a) history (or family history) of seizure or epilepsy; b) history of stroke, head injury, or unexplained seizures; c) concurrent medication use such as tricyclic antidepressants, neuroleptic medications, or other drugs that are known to lower the seizure threshold; d) secondary conditions that may significantly alter electrolyte balance or lower seizure threshold; e) no quantifiable motor threshold such that TMS dosage cannot be accurately determined.
11. Known bee, insect, or arachnid allergy
12. Other medical contraindications to any of the study procedures.

Participants will be assigned course credit or receive financial compensation after participating in the study. Those who participate through SONA recruitment will receive course credit. Participants will sign up for the study only if they are able to make all four visits of the experiment. If a participant does not attend all three visits, course credit will still be given for the amount of time the participant spent doing the experiment (i.e., 1 credit for 1 hour).

After screening, participants will be emailed blank copies of the forms, questionnaires, and screening tools that will be completed during the first visit, and they will be informed that they may complete the forms in advance and bring the completed forms with them to save time, should they desire. They will be asked to not return their forms via email, and to only bring them to the first visit.

DAY 1 On Day 1, participants will first provide informed consent after the nature of the study has been fully explained and the participant has had time to ask questions. After obtaining informed consent, participants will complete a demographics and eligibility questionnaire (see Section 10.1, Item 1.0) or hand in their already-completed forms, which will be reviewed by the researcher upon completion. Ineligible participants (i.e., participants with bee, insect, or spider allergies, with scores below 17 on the SPQ, who do not speak English, are taking medications that lower the seizure threshold, or other exclusion criteria as listed in section 11.1) will be informed that they do not meet criteria and the research session will be terminated at this time. Participants found to be ineligible will still receive 1 credit for their time. All to-be-administered questionnaires are listed below and uploaded in Section 10.1, Item 1.0 of this IRB submission.

Spider Phobia Questionnaire (SPQ; Klorman et al, 1974) Demographics & Eligibility Questionnaire Fear of Spiders Questionnaire (FSQ; Szymanski & O'Donohue, 1995) PHQ2 PHQ9 Hamilton Rating Scale for Depression (specifically the suicidality item) GAD7 Tracking and Reimbursement (this questionnaire is used exclusively to track the number of visits completed and information necessary to ensuring that participants receive the proper financial or course credit compensation for their time; it contains no research data used for the study)

All participants will complete a BAT with a live tarantula. This phase of the experiment consists of 9 steps, lasting 30 seconds each with a 30 second pause between each step. During the BAT, self-reported and physiological data will be collected at each step. Skin conductance response (SCR) and heart-rate variability (HRV) will be utilized as physiologic measures of fearful arousal using BIOPAC MP150 hardware and AcqKnowledge version 4.2 software (BIOPAC Systems, Inc.).(Appelhans & Luecken, 2006; Choi et al., 2017; Christopoulos, Uy, & Yap, 2016; Laine, Spitler, Mosher, & Gothard, 2009; Thayer, Åhs, Fredrikson, Sollers, & Wager, 2012; Williams et al., 2001) Baseline SCR and HRV will be measured during a 3-minute prior to initiation of a BAT. SCR will be recorded from electrodes attached to the subjects' second and third fingers. Average SCRs and peak SCRs at each step will be measured and compared to individual baselines. HRV will be calculated from R-R intervals in a lead II electrode configuration recording; average HRVs from each step will be compared to individual baselines. The steps are as follows:

1. Stand 5 feet away from tarantula in closed terrarium
2. Stand 1 foot away from tarantula in terrarium with top removed
3. Place both hands on the side of terrarium with top removed
4. Touch nose against the glass of terrarium while looking at the tarantula
5. Place gloved hand halfway inside terrarium
6. Place gloved hand inside terrarium with all fingertips touching base of terrarium
7. Place bare hand inside terrarium with all fingertips touching base of terrarium
8. Touch the back of the tarantula's leg continuously with a Q-tip
9. Touch the back of the tarantula's leg continuously with the tip of the index finger

Prior to beginning the BAT, all participants will be read instructions reporting the following: The experiment consists of 9 steps, each lasting 30 seconds. Instructions for each step will be read aloud before the participant proceed to the next step. Each step must be completed before moving on to the next step, and steps much be completed in sequential order. During each step, participant's heart rate and sweating will be recorded via the electrodes on participant's chest and finger. After the experimenter reads the instructions for the next step and prior to completing the step, the participant will also be asked to rate participant's confidence level to complete the step on a scale from 0 to 100 (0= no confidence, 25= mild confidence, 50= moderate confidence, 75= high confidence, 100 = complete confidence) and participant's anticipatory distress on a scale from 0 to 100 (0=no distress, 25=mild distress, 50=moderate distress, 75= high distress, 100= severe distress). After completion of each step, participants will be asked to rate their maximum level of distress during the step on a scale from 0 to 100. Participants are entitled to withdraw at any step if they do not wish to continue. At this point participants will have an opportunity to ask questions before beginning testing. The first step of the experiment is to stand 5 feet away from the tarantula while it is in its closed container for 30 seconds. The final step of the experiment is to touch the back of the tarantula's leg with the tip of participant's index finger continuously for 30 seconds.

Before beginning the BAT and after ensuring comprehension of the above instructions, the experimenter will ask the participant to rate his/her overall confidence and overall anticipatory distress with respect to his/her ability to complete all nine steps (see rating scales in above instructions). Before each subsequent step, the participant will be asked to rate his/her confidence and anticipatory distress regarding his/her ability to complete that particular step. During each step, the experimenter will record the spider's movement on a categorical scale (0 = no movement, 1 = a little movement, 2 = a lot of movement). After each step, the participant will be asked to rate his/her maximum level of distress while completing that particular step. Finally, the experimenter will record the number of steps willingly completed for a given participant.

Next, all participants will engage in a series of exposure practices with a different live tarantula from the one they saw during the BAT. Exposure therapy will consist of a series of 10 identical exposure trials of a 30-second duration with a 30-second pause between trials. Participants will be asked to place an ungloved hand in the terrarium (with all fingertips touching the base of the terrarium) on the opposite end of the terrarium as the tarantula during the trial. Prior to completing the series of exposures, participants will be asked about their feared outcome concerning approaching the tarantula (e.g., being bitten). Participants are entitled to withdraw at any step during exposures and will not be prevented from further continuation in the study.

Following the series of exposures, participants will undergo TMS treatments using an iTBS protocol. Before the first iTBS treatment, the TMS coil will be calibrated to the subject's individual resting motor threshold (RMT), or the minimum stimulus intensity necessary to elicit a motor response in the right abductor pollicis brevis (APB) or first dorsal interosseus (FDI) muscles for ≥ 50% of stimuli applied to the motor cortex. After initial calibration, the TMS coil will be placed over the subject's ventral medial prefrontal cortex (vmPFC; as determined using position Fpz of the international 10-20 EEG electrode system), a TMS target shown to affect phobic response.(Baeken et al., 2010; Guhn et al., 2012, 2014; Suarez-Jimenez et al., 2018) Stimulation intensity of 100% of the individual RMT in bursts of three pulses at a frequency of 50 Hz every 200 ms on top of a 5Hz carrier wave. Pulse delivery is over 2 s and repeated every 10 s, 20 times in succession, for a total of 600 pulses delivered in 3.33 minutes.(Baeken et al., 2010; Bulteau et al., 2017; Guhn et al., 2014) This specific protocol was selected based on the assumption that it should impact fear circuitry top-down from prefrontal to subcortical networks (particularly the amygdala) as seen in prior work.(Baeken et al., 2010; Bulteau et al., 2017; Guhn et al., 2014) Control iTBS will consist of the same stimulation parameters over the subject's midline central sulcus or vertex (as determined using position Cz, of the international 10-20 EEG electrode system). This placement was chosen for control as its position over the vertex will minimize amount of cortex stimulated and the stimulated area is not associated with the circuitry examined in this experiment.(Duecker & Sack, 2015) It is a commonly-used control site in TMS studies because it is associated with no known effects and has a similar risk profile to other TMS sites. (Foltys et al., 2001; Jung, Bungert, Bowtell, & Jackson, 2016; Rossi et al., 2009; Weiss, Sparing, Fink, Tomasino, & Dafotakis, 2008) It is generally associated with lower rates of scalp discomfort and no clinically-observed behavioral or mood effects.(Jung et al., 2016; Rossi et al., 2009) Some work has demonstrated a possible decrease in activation of the default mode network, though this has not been found to be clinically-significant.(Jung et al., 2016)

DAY 2 As described above, this visit will occur one to two days after Day 1. All participants will return to the laboratory to engage in a second series of exposure practices with the same tarantula from exposures at the first visit. They will undergo 10 identical exposure trials for durations of 30 seconds each, with a 30-second pause between trials. During each exposure trial, they will again be asked to place an ungloved hand in the terrarium (with all fingertips touching the base of the terrarium) on the opposite end of the terrarium as the tarantula during the trial. Prior to completing the series of exposures, participants will be asked about their feared outcome concerning approaching the tarantula (e.g., being bitten). Participants are entitled to withdraw at any step during exposures and will not be prevented from further continuation in the study.

Following the series of exposure practices, participants will undergo a TMS treatment using an iTBS treatment protocol in the same location that they received stimulation on Day 1 (vmPFC vs. vertex).

DAY 3 This visit will be identical to Day 2, and will occur one to two days after Day 2.

DAY 4 This visit will occur five to seven days after Day 3. All participants will complete the Spider Phobia Questionnaire (SPQ; Klorman et al, 1974) and Fear of Spiders Questionnaire (FSQ; Szymanski & O'Donohue, 1995), uploaded in Section 10.1, Item 1.0, to test for change in arachnophobia fear/avoidance symptoms as a function of TMS treatment received. Next, all participants will complete an identical BAT to that completed at their first visit with the same tarantula (see DAY 1 above). Self-report and physiological (i.e., SCR) data will again be collected. After completion of these forms, participants will be debriefed by an un-blinded member of the study team and informed to which group they are assigned. They will be encouraged to discuss whatever questions or concerns they have regarding the study at that time.

After completion of Day 4, participants will be compensated for their time with one credit per hour of study participation.

Dependent variables (DVs) will be quantitative self-reports and behavioral symptoms of fear and avoidance of spiders both pre- and post-treatment, including SCR (difference between baseline and average level during BAT anticipation period, and number of peaks during BAT), total number of steps completed during the BAT, self-reported distress, anticipatory distress, and maximum distress per BAT step, and total score on the SPQ. BAT measures will be collected for each step and therefore minima, maxima, and means will be compared between the two groups. Primary outcomes examined will be number of steps completed during BAT, self-reported distress during BAT, number of SCR peaks during BAT, SPQ score, and FOS score. All other variables examined will be secondary outcomes. Additionally, for feasibility and tolerability assessment, attendance to TMS treatment sessions and early termination of TMS treatment sessions will be recorded. The primary independent variable examined will be the treatment group (iTBS vs. control iTBS). The sample size will be 40 participants (20 per group). Pre-comparison ANOVA will be performed to limit type 1 error due to multiplicity of comparisons.

Hypotheses will be tested using between-group two-tailed t-tests given that investigators are testing not only for magnitude of an effect, but also direction of an effect. Investigators expect that comparisons of efficacy will demonstrate increased confidence during BAT approach, decreased endorsed fear of spiders as measured by SPQ and FSQ, and reduced physiologic response to stimulus (reduced HRV and SCR) with active iTBS and exposure when compared to control iTBS and exposure. Investigators expect that comparisons of feasibility and tolerability will show no significant difference between attendance to, early termination of, or subjective tolerability ratings of TMS treatment sessions between treatment groups.

ADVERSE EVENT MANAGEMENT Study personnel administering the BAT and exposure treatments will be bachelors-level trained or current UCLA students. These personnel have not been identified at this time, but will be added to the IRB and protocols as they are identified. They will be trained by personnel from Anxiety and Depression Research Center (ADRC; personnel under the supervision of Dr. Michelle Craske) in both how to properly administer the BAT and exposure treatments, as well as how to address any questions, concerns, or unexpected events that arise from these treatments (including acute episodes of psychological distress, escape of spiders, etc.). These personnel have ample experience in training others how to administer these treatments.

Three Chilean Rose Tarantulas (Grammostola rosea) will be stored in individual terrariums with weighted lids in a locked room within the ADRC (Life Sciences 5347), under the supervision of Dr. Michelle Craske and her laboratory personnel. All BATs and exposure treatments will take place in a controlled closed room without windows, open vents, or other large openings, to minimize the likelihood of a tarantula escape. At the beginning and end of every study session, study personnel will confirm the presence of the tarantula within the terrarium and confirm complete closure of the terrarium. After termination of testing for the day, study personnel will again confirm of the presence of the spider and the terrarium closure before departing.

In the event that a spider should escape from its terrarium, the participant will be removed from the room and study personnel will immediately re-close the room, search for the tarantula, and transfer it back to the terrarium in a manner safe for both the personnel and the spider when found. This will involve coaxing the spider to a sealable pre-dampened carrier, temporarily sealing it, and opening it inside the spider's terrarium. Though the risk posed by a tarantula bite or hair projection is low and the risk of occurrence is low, study personnel will don gloves, eye protection, and a long-sleeved labcoat (all three of which will be provided) before attempting transfer to minimize this risk. If not found after a thorough search, the room will remain closed, and other laboratory personnel and the PI will be notified, and further action will be taken to locate the spider.

Any injury sustained in the process of a spider escape or containment, such as a spider bite, will be reported as an adverse event. Should such an event emerge, study personnel present at the time of the event will be asked to contact the PI or a study clinician, who will assess the severity of the event. If the PI is not contacted in real-time, personnel will contact the PI within 24 hours of the event, and the PI will then report the adverse event within 24 hours of being informed.

Investigators will employ the following strategy to manage suicidality and other serious adverse events (SAEs). All exposure and TMS procedures will be performed during normal working hours while there is a psychiatrist on duty at the Clinical TMS Service. Should participants become acutely distressed during a study visit, the attending psychiatrist on duty will take any steps necessary to address any clinical issues that emerge. The PI will follow up with all participants by phone 12-24 hours after all exposure treatments to ensure that they are not suffering from ongoing distress, and participants will be given contact information for the PI to reach out sooner should they desire. The PI will involve licensed clinicians as appropriate. At the initial study visit, subjects will complete the PHQ2 (reflex to PHQ9), GAD7, and HamD suicidality item and review their responses with a research assistant and clinician. All subjects also will be reminded at each visit about the availability of a clinician should the subject develop any event of concern, including suicidality or adverse events. Should such an event emerge, the subject will be instructed to contact the PI or a study clinician, who will assess the presentation as per their standard clinical protocol. This assessment will categorize the SAE as emergent or nonemergent. For non-emergent events, the clinicians will manage as they see fit. Rapid consultation with the Principal Investigator is available; should the clinician contact the PI, he or she will then be responsible for reporting the event as an SAE. If a consultation with the PI is not pursued in real-time, the clinician will inform the PI of the event within 24 hours of having identified the event. For emergent events, such as the worsening of suicidality or self-injurious behavior, the clinician will instruct the subject to go to the nearest emergency room possible. Should the clinician be concerned about the subject's imminent safety, he or she may contact the individual named by the subject in the consent form as the emergency contact, so that the contact person may help the subject get to an emergency room. If such an action is not feasible, the clinician may petition the subject to be brought involuntarily to the nearest emergency room possible, as provided for under state mental health laws in California where the study is being conducted. Consultation at any time is available by contacting the PI or a study clinician. Should the PI be contacted in real-time, he will then be responsible for initiating the SAE reporting. If the PI is not contacted in real-time, the clinician will contact the PI within 24 hours of the event, and the PI will then complete SAE reporting within 24 hours of being informed. All reports of adverse events will be reviewed by the PI and reported to the UCLA Institutional Review Board in accordance with its policies.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. English-speaking
3. Spider phobia as determined by a Spider Phobia Questionnaire (SPQ; Klorman et al 1974) score of at least 17/30

Exclusion Criteria:

1. Subject is mentally or legally incapacitated, unable to give informed consent.
2. Subjects with psychosis (psychotic depression, schizophrenia, or schizoaffective diagnoses (lifetime)); bipolar disorder (lifetime); dementia (lifetime); delirium within the past 6 months; eating disorder within the past year; obsessive-compulsive disorder (lifetime); post-traumatic stress disorder within the past year; acute risk for suicide or self-injurious behavior. Patients with diagnostic uncertainty or ambiguity (e.g. rule-out pseudodementia of depression) will be excluded.
3. Subjects with a HamD suicidality item score of '3' or '4,' corresponding to "suicidal ideas or gestures" or "attempts at suicide," will be excluded.
4. Subjects with exposure to ECT within the past 6 months, previous TMS treatment for any condition, or VNS treatment (lifetime).
5. Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke, CVA, or TIAs; cerebral aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.
6. Any history of intracranial implant including cochlear implant, implanted electrodes/stimulators, aneursym clips or coils, stents, bullet fragments; implanted cardiac pacemaker, defibrillator, vagus nerve stimulator, deep brain stimulator; or other implanted devices or objects contraindicated by product labeling.
7. Neurological conditions including epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, history of repetitive or severe head trauma, or with primary or secondary tumors in the CNS.
8. current pregnancy or breast feeding. The effects of TMS on pregnant and breastfeeding patients has not been systematically studied.
9. Infection or loss of integrity of skin over the forehead, where the device will be positioned.
10. Increased risk of seizure as indicated by: a) history (or family history) of seizure or epilepsy; b) history of stroke, head injury, or unexplained seizures; c) concurrent medication use such as tricyclic antidepressants, neuroleptic medications, or other drugs that are known to lower the seizure threshold; d) secondary conditions that may significantly alter electrolyte balance or lower seizure threshold; e) no quantifiable motor threshold such that TMS dosage cannot be accurately determined.
11. Known bee, insect, or arachnid allergy
12. Other medical contraindications to any of the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Leuchter, B.S., Principal Investigator — University of California, Los Angeles; Marco Iacoboni, M.D., Ph.D., Principal Investigator — Professor, UCLA Psychiatry and Biobehavioral Science
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appelhans, B. M., & Luecken, L. J. (2006). Heart rate variability as an index of regulated emotional responding. Review of General Psychology, 10(3), 229-240. http://doi.org/10.1037/1089-2680.10.3.229
- [Background] Baeken C, De Raedt R, Van Schuerbeek P, Vanderhasselt MA, De Mey J, Bossuyt A, Luypaert R. Right prefrontal HF-rTMS attenuates right amygdala processing of negatively valenced emotional stimuli in healthy females. Behav Brain Res. 2010 Dec 25;214(2):450-5. doi: 10.1016/j.bbr.2010.06.029. Epub 2010 Jul 1. PMID 20600336
- [Background] Bulteau S, Sebille V, Fayet G, Thomas-Ollivier V, Deschamps T, Bonnin-Rivalland A, Laforgue E, Pichot A, Valriviere P, Auffray-Calvier E, Fortin J, Pereon Y, Vanelle JM, Sauvaget A. Efficacy of intermittent Theta Burst Stimulation (iTBS) and 10-Hz high-frequency repetitive transcranial magnetic stimulation (rTMS) in treatment-resistant unipolar depression: study protocol for a randomised controlled trial. Trials. 2017 Jan 13;18(1):17. doi: 10.1186/s13063-016-1764-8. PMID 28086851
- [Background] Choi KH, Kim J, Kwon OS, Kim MJ, Ryu YH, Park JE. Is heart rate variability (HRV) an adequate tool for evaluating human emotions? - A focus on the use of the International Affective Picture System (IAPS). Psychiatry Res. 2017 May;251:192-196. doi: 10.1016/j.psychres.2017.02.025. Epub 2017 Feb 11. PMID 28213189
- [Background] Christopoulos, G. I., Uy, M. A., & Yap, W. J. (2016). The Body and the Brain: Measuring Skin Conductance Responses to Understand the Emotional Experience. Organizational Research Methods, 1-27. http://doi.org/10.1177/1094428116681073
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Demitrack MA, Thase ME. Clinical significance of transcranial magnetic stimulation (TMS) in the treatment of pharmacoresistant depression: synthesis of recent data. Psychopharmacol Bull. 2009;42(2):5-38. PMID 19629020
- [Background] Deppermann S, Notzon S, Kroczek A, Rosenbaum D, Haeussinger FB, Diemer J, Domschke K, Fallgatter AJ, Ehlis AC, Zwanzger P. Functional co-activation within the prefrontal cortex supports the maintenance of behavioural performance in fear-relevant situations before an iTBS modulated virtual reality challenge in participants with spider phobia. Behav Brain Res. 2016 Jul 1;307:208-17. doi: 10.1016/j.bbr.2016.03.028. Epub 2016 Mar 17. PMID 26996315
- [Background] Duecker F, Sack AT. Rethinking the role of sham TMS. Front Psychol. 2015 Feb 26;6:210. doi: 10.3389/fpsyg.2015.00210. eCollection 2015. PMID 25767458
- [Background] Foltys H, Sparing R, Boroojerdi B, Krings T, Meister IG, Mottaghy FM, Topper R. Motor control in simple bimanual movements: a transcranial magnetic stimulation and reaction time study. Clin Neurophysiol. 2001 Feb;112(2):265-74. doi: 10.1016/s1388-2457(00)00539-3. PMID 11165528
- [Background] Guhn A, Dresler T, Andreatta M, Muller LD, Hahn T, Tupak SV, Polak T, Deckert J, Herrmann MJ. Medial prefrontal cortex stimulation modulates the processing of conditioned fear. Front Behav Neurosci. 2014 Feb 18;8:44. doi: 10.3389/fnbeh.2014.00044. eCollection 2014. PMID 24600362
- [Background] Guhn A, Dresler T, Hahn T, Muhlberger A, Strohle A, Deckert J, Herrmann MJ. Medial prefrontal cortex activity during the extinction of conditioned fear: an investigation using functional near-infrared spectroscopy. Neuropsychobiology. 2012 Jun;65(4):173-82. doi: 10.1159/000337002. Epub 2012 Apr 26. PMID 22538209
- [Background] Jung J, Bungert A, Bowtell R, Jackson SR. Vertex Stimulation as a Control Site for Transcranial Magnetic Stimulation: A Concurrent TMS/fMRI Study. Brain Stimul. 2016 Jan-Feb;9(1):58-64. doi: 10.1016/j.brs.2015.09.008. Epub 2015 Sep 25. PMID 26508284
- [Background] Klorman, R., Weerts, T. C., Hastings, J. E., Melamed, B. G., & Lang, P. J. (1974). Psychometric description of some specific-fear questionnaires. Behavior Therapy, 5(3), 401-409. http://doi.org/10.1016/S0005-7894(74)80008-0
- [Background] Laine CM, Spitler KM, Mosher CP, Gothard KM. Behavioral triggers of skin conductance responses and their neural correlates in the primate amygdala. J Neurophysiol. 2009 Apr;101(4):1749-54. doi: 10.1152/jn.91110.2008. Epub 2009 Jan 14. PMID 19144740
- [Background] Leuchter AF, Hunter AM, Krantz DE, Cook IA. Rhythms and blues: modulation of oscillatory synchrony and the mechanism of action of antidepressant treatments. Ann N Y Acad Sci. 2015 May;1344(1):78-91. doi: 10.1111/nyas.12742. Epub 2015 Mar 23. PMID 25809789
- [Background] Mutz J, Edgcumbe DR, Brunoni AR, Fu CHY. Efficacy and acceptability of non-invasive brain stimulation for the treatment of adult unipolar and bipolar depression: A systematic review and meta-analysis of randomised sham-controlled trials. Neurosci Biobehav Rev. 2018 Sep;92:291-303. doi: 10.1016/j.neubiorev.2018.05.015. Epub 2018 May 12. PMID 29763711
- [Background] Notzon S, Deppermann S, Fallgatter A, Diemer J, Kroczek A, Domschke K, Zwanzger P, Ehlis AC. Psychophysiological effects of an iTBS modulated virtual reality challenge including participants with spider phobia. Biol Psychol. 2015 Dec;112:66-76. doi: 10.1016/j.biopsycho.2015.10.003. Epub 2015 Oct 22. PMID 26476332
- [Background] Paes F, Baczynski T, Novaes F, Marinho T, Arias-Carrion O, Budde H, Sack AT, Huston JP, Almada LF, Carta M, Silva AC, Nardi AE, Machado S. Repetitive Transcranial Magnetic Stimulation (rTMS) to Treat Social Anxiety Disorder: Case Reports and a Review of the Literature. Clin Pract Epidemiol Ment Health. 2013 Oct 31;9:180-8. doi: 10.2174/1745017901309010180. eCollection 2013. PMID 24278088
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Suarez-Jimenez B, Bisby JA, Horner AJ, King JA, Pine DS, Burgess N. Linked networks for learning and expressing location-specific threat. Proc Natl Acad Sci U S A. 2018 Jan 30;115(5):E1032-E1040. doi: 10.1073/pnas.1714691115. Epub 2018 Jan 11. PMID 29326231
- [Background] Szymanski J, O'Donohue W. Fear of Spiders Questionnaire. J Behav Ther Exp Psychiatry. 1995 Mar;26(1):31-4. doi: 10.1016/0005-7916(94)00072-t. PMID 7642758
- [Background] Thayer JF, Ahs F, Fredrikson M, Sollers JJ 3rd, Wager TD. A meta-analysis of heart rate variability and neuroimaging studies: implications for heart rate variability as a marker of stress and health. Neurosci Biobehav Rev. 2012 Feb;36(2):747-56. doi: 10.1016/j.neubiorev.2011.11.009. Epub 2011 Dec 8. PMID 22178086
- [Background] Williams LM, Phillips ML, Brammer MJ, Skerrett D, Lagopoulos J, Rennie C, Bahramali H, Olivieri G, David AS, Peduto A, Gordon E. Arousal dissociates amygdala and hippocampal fear responses: evidence from simultaneous fMRI and skin conductance recording. Neuroimage. 2001 Nov;14(5):1070-9. doi: 10.1006/nimg.2001.0904. PMID 11697938
- [Background] Tomasino B, Fink GR, Sparing R, Dafotakis M, Weiss PH. Action verbs and the primary motor cortex: a comparative TMS study of silent reading, frequency judgments, and motor imagery. Neuropsychologia. 2008;46(7):1915-26. doi: 10.1016/j.neuropsychologia.2008.01.015. Epub 2008 Feb 2. PMID 18328510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 8/2019 to 3/2020. Study ended early due to COVID restrictions, as well as personnel and equipment limitations.
Groups:
- Active iTBS, Ventromedial Prefrontal Cortex (vmPFC): Stimulation intensity of 100% of the individual resting motor threshold in bursts of three pulses at a frequency of 50 Hz every 200 ms on top of a 5Hz carrier wave. Pulse delivery is over 2 s and repeated every 10 s, 20 times in succession, for a total of 600 pulses delivered in 3.33 minutes.
  Delivered over vmPFC, as determined by position Fpz of the international 10-20 EEG electrode system.
  Intermittent Theta Burst Stimulation (iTBS), Ventromedial Prefrontal Cortex (vmPFC): iTBS delivered to vmPFC for active treatment of spider phobia.
- Control iTBS, Vertex: Stimulation intensity of 100% of the individual resting motor threshold in bursts of three pulses at a frequency of 50 Hz every 200 ms on top of a 5Hz carrier wave. Pulse delivery is over 2 s and repeated every 10 s, 20 times in succession, for a total of 600 pulses delivered in 3.33 minutes.
  Delivered over vertex, as determined by position Cz of the international 10-20 EEG electrode system.
  Intermittent Theta Burst Stimulation (iTBS), vertex: iTBS delivered to vertex for placebo treatment of spider phobia.
Period: Overall Study
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Started | 11 | 11
Completed | 8 | 9
Not Completed | 3 | 2
Not completed — Inadvertent Enrollment, discovered to meet exclusion criteria after enrollment | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (2.3) | 21 (3.8) | 21 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 1 | 5 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 17
Patient Health Questionnaire (PHQ-9) score [Mean (Standard Deviation); unit: units on a scale] — Baseline score on PHQ9. Utilized as a screening tool to reduce likelihood of enrollment with co-morbid depression. Scored from 0 to 27, with a higher score indicating a higher burden of depression.
  units on a scale | 2.11 (1.67) | 1.91 (1.70) | 2.00 (1.62)
Generalized Anxiety Disorder 7 (GAD7) questionnaire [Mean (Standard Deviation); unit: units on a scale] — GAD7 questionnaire score utilized as a screening tool for those with anxiety disorders other than specific phobia. Scored from 0 to 21, with higher scores indicating a greater burden of anxiety.
  units on a scale | 3.22 (2.83) | 2.55 (2.02) | 2.85 (2.35)

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Approach Test, Change in Steps Completed
Description: The difference between the number of steps completed during the pre- and post-treatment behavioral approach tests.
Time Frame: baseline and 1 week after treatment
Measure: Mean (Standard Error); unit: Steps
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
Steps | 0 (0.19) | 0.78 (0.33)
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Test type: Superiority — Repeated-measure MANOVA was utilized to compare control and active group; p = 0.518, ANOVA

2. Primary Outcome: Change in Subjective Distress, Klorman Spider Phobia Questionnaire
Description: Changes in scores on questionnaires regarding distress around spiders (Klorman spider phobia questionnaire). Scored on a scale of 0-31, with higher numbers associated with greater subjective fear of spiders. No subscales reported
Time Frame: baseline and 1 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
score on a scale | 4.25 (0.73) | 4.56 (0.66)
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Test type: Superiority — Repeated-measure MANOVA was utilized to compare control and active group. This allowed for examination between and within each group. Analysis described here is within-group differences; p = 0.008, ANOVA — a priori threshold for significance of p=0.05. Observed power η2=0.39
Statistical Analysis 2: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Test type: Superiority — Repeated-measure MANOVA was utilized to compare control and active group. This allowed for examination between and within each group. Analysis described here is between-group differences; p > 0.05, ANOVA — a priori threshold for significance of p=0.05

3. Primary Outcome: Change in Subjective Distress, Syzmanski Fear of Spiders Questionnaire
Description: Changes in scores on questionnaires regarding distress around spiders (Syzmanski Fear of Spiders Questionnaire). 18 items each scored on a scale of 1-7 (total score ranging 18-126), with higher numbers associated with greater subjective fear of spiders. No subscales reported
Time Frame: baseline and 1 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
score on a scale | 22.75 (3.92) | 16.67 (1.65)
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Test type: Superiority — Repeated-measure MANOVA was utilized to compare control and active group. This allowed for examination between and within each group. Result described here is within-group difference over time; p = 0.004, ANOVA — a priori threshold for significance p=0.05. Result above describes within group testing over time. Observed power η2=0.43
Statistical Analysis 2: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Test type: Superiority — Repeated-measure MANOVA was utilized to compare control and active group. This allowed for examination between and within each group. Result described here is the between-group comparison; p > 0.05, ANOVA — a priori threshold for significance p=0.05

4. Secondary Outcome: Behavioral Approach Test, Change in Skin Conductance
Description: The difference between the change in skin conductance measured during each step of the pre- and post-treatment behavioral approach tests (BATs). Differences were only compared in steps that subjects completed during both pre- and post-treatment BATs.
Time Frame: baseline and 1 week after treatment
Population: One subject within the active group was noted to have corrupted skin conductance data during analysis of post-treatment data and thus that subject's physiologic data was unable to be used for SCL analysis.Per Behavioral Approach Test (BAT) protocol, the test was ended when subjects were unable to complete a step. The number analyzed at each step reflects the number of subjects who completed that step in that group both before and after treatment.
Measure: Mean (Standard Error); unit: micro-siemens
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 7 | 9
micro-siemens
  Step 1 | .27 (1.67) | 4.75 (2.48)
  Step 2 | -0.36 (1.20) | 4.79 (2.30)
  Step 3 | -0.11 (1.17) | 4.70 (2.56)
  Step 4: number analyzed (Participants) | 7 | 8
  Step 4 | -0.51 (1.43) | 4.65 (2.54)
  Step 5: number analyzed (Participants) | 6 | 6
  Step 5 | -0.16 (1.67) | 5.50 (3.19)
  Step 6: number analyzed (Participants) | 5 | 5
  Step 6 | -0.59 (1.64) | 0.74 (0.91)
  Step 7: number analyzed (Participants) | 4 | 3
  Step 7 | -1.65 (1.90) | 2.61 (1.30)
  Step 8: number analyzed (Participants) | 2 | 1
  Step 8 | -1.87 (1.03) | -0.27 (NA) — Single data point, no standard error available
  Step 9: number analyzed (Participants) | 1 | 0
  Step 9 | -0.9 (NA) — Single data point, no standard error available |
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Goodness of fit test of a two-variable negative binomial multi-level model of skin conductance level (SCL) as a function of step and timepoint. This multi-level model was generated using the menbreg function in Stata 16; Test type: Other — This was a goodness of fit test of a multi-level model, fit was tested using a wald chi-square test; p < 0.01, Chi-squared — Threshold for significance was p=0.05; This was specifically a wald chi-square test, performed in Stata for the purpose of assessing goodness-of-fit of a mixed effects model
Statistical Analysis 2: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; The second statistical analysis involved testing of the step-by-timepoint interaction in the two-variable negative binomial model of skin conductance level (SCL) (as a function of step and timepoint); Test type: Superiority; p = 0.029, Mixed Models Analysis — a priori threshold for significance of 0.05

5. Secondary Outcome: Change in Subjective Anticipatory Distress, Behavioral Approach Test
Description: Changes in subjective pre-step anticipatory distress (reported 0-100) reported prior to each step during the behavioral approach test. Positive score indicates corresponding reduction in distress from pre- to post-treatment.
Time Frame: baseline and 1 week, difference reported
Population: Per Behavioral Approach Test (BAT) protocol, the test was ended when subjects were unable to complete a step. The number analyzed at each step reflects the number of subjects who completed that step in that group both before and after treatment, and compares the subject's data from before to after treatment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
score on a scale
  Step 1 | 0.57 (7.47) | 26.89 (9.01)
  Step 2 | 4.86 (14.43) | 35.56 (7.42)
  Step 3 | 11.86 (12.09) | 39.44 (6.64)
  Step 4: number analyzed (Participants) | 8 | 8
  Step 4 | 17.57 (11.27) | 41.25 (6.60)
  Step 5: number analyzed (Participants) | 7 | 6
  Step 5 | 12.33 (7.92) | 45.83 (6.76)
  Step 6: number analyzed (Participants) | 7 | 5
  Step 6 | 16.0 (7.97) | 42.0 (11.58)
  Step 7: number analyzed (Participants) | 6 | 3
  Step 7 | 16.25 (7.42) | 48.3 (12.02)
  Step 8: number analyzed (Participants) | 4 | 1
  Step 8 | 17.5 (2.50) | 10.0 (NA) — Single data point, no standard error available
  Step 9: number analyzed (Participants) | 1 | 0
  Step 9 | 10.0 (NA) — Single data point, no standard error available |
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Goodness of fit test of a two-variable negative binomial multi-level model of anticipatory distress as a function of step and timepoint. This multi-level model was generated using the menbreg function in Stata 16; Test type: Other — This was a goodness of fit test of a multi-level model, fit was tested using a wald chi-square test; p < 0.001, Chi-squared — a priori threshold for significance was p=0.05; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; This statistical analysis involved testing of the step-by-timepoint interaction in the two-variable negative binomial model of anticipatory distress as a function of step and timepoint; Test type: Superiority; p = 0.63, Mixed Models Analysis — a priori threshold for significance of 0.05
Statistical Analysis 3: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Goodness of fit test of a two-variable negative binomial multi-level model of anticipatory distress as a function of treatment group and timepoint. This multi-level model was generated using the menbreg function in Stata 16; Test type: Other — This was a goodness of fit test of a multi-level model, fit was tested using a wald chi-square test; p < .001, Chi-squared — a priori threshold for significance of p=0.05; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; This statistical analysis involved testing of the step-by-timepoint interaction in the two-variable negative binomial model of anticipatory distress as a function of group and timepoint; Test type: Superiority; p < 0.001, Mixed Models Analysis — a priori threshold for significance of 0.05
Statistical Analysis 5: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Goodness of fit test of a two-variable negative binomial multi-level model of anticipatory distress as a function of step and group. This multi-level model was generated using the menbreg function in Stata 16; Test type: Other — This was a goodness of fit test of a multi-level model, fit was tested using a wald chi-square test; p < 0.001, Chi-squared — a priori threshold for significance was p=0.05; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; This statistical analysis involved testing of the step-by-timepoint interaction in the two-variable negative binomial model of anticipatory distress as a function of step and group; Test type: Superiority; p = 0.047, Mixed Models Analysis — a priori threshold for significance of 0.05

6. Secondary Outcome: Average Treatment Intensity Tolerated
Description: The TMS treatment intensity tolerated by subjects in each group, averaged over the 3-day course of treatment for each subject. Ranges from 80-100% and is defined in reference to the subject's motor threshold.
Time Frame: Average tolerated intensity during TMS treatment sessions (days 1, 2, and 3 of treatment)
Measure: Mean (Standard Error); unit: percentage of motor threshold
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
percentage of motor threshold | 90.8 (2.87) | 98.8 (0.85)
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; 2-sided Mann-Whitney U Test (nonparametric) utilized to compare the ability of the groups to tolerate treatment intensity; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney) — a priori threshold for significance of p=0.05; Mann Whitney U statistic = 13.5, Standard Error of Mean 9.58

7. Other Pre Specified Outcome: Pain Score
Description: The average post-treatment pain score as defined by the short-form 15-item McGill pain scale (scored from 0 to 45, with a higher score indicating a greater degree of pain, and a lower score indicating less pain). Each individual subject's average score was calculated by averaging his/her respective scores collected after each of the three TMS sessions. Each group's average score was calculated by averaging the average pain scores of each subject.
Time Frame: Days 1, 2, and 3 (after each TMS treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
score on a scale | 3.33 (1.47) | 1.67 (0.64)

8. Other Pre Specified Outcome: Group Assignment Conjecture
Description: After completion of all other study-related activities and questionnaires (i.e. after completing post-treatment SPQ, FOS, and BAT during the followup visit), subjects were asked to guess to which group they had been assigned after completing the study and before being unblinded by the PI. Raters were also asked to guess to which group each subject had been assigned. Chi-squared analyses were performed for both subjects and raters for each group to validate blinding.
Time Frame: Immediately following repeat behavioral approach testing (i.e. the very last activity of the final/4th/followup visit).
Measure: Number; unit: guesses
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
guesses
  Number of correct subject guesses | 5 | 4
  Number of correct rater guesses | 4 | 5
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Test type: Other — A pair of chi-square analyses were performed to validate blinding of the study (based on questionnaires completed by subjects and raters). Given the small sample size, Fisher's exact method was utilized. The number of correct and incorrect guesses for each group were examined once for the subject guesses and once for the rater's guesses; p > .05, Fisher Exact; For the subjects, p=0.64 using Fisher's exact method. For the raters, p=1 using Fisher's exact method

9. Secondary Outcome: Change in Subjective Maximum Distress, Behavioral Approach Test
Description: Changes in subjective post-step maximum distress (reported 0-100) reported immediately following each step during the behavioral approach test. Positive change in score represents a corresponding reduction in relative distress.
Time Frame: baseline and 1 week, change in scores from pre to post reported
Population: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
Number analyzed (Participants) | 8 | 9
score on a scale
  Step 1 | -5.14 (6.02) | 18.33 (7.78)
  Step 2 | 10.43 (11.31) | 32.78 (8.58)
  Step 3 | 10.43 (13.04) | 38.33 (6.92)
  Step 4: number analyzed (Participants) | 8 | 8
  Step 4 | 13.83 (14.93) | 28.13 (9.86)
  Step 5: number analyzed (Participants) | 7 | 6
  Step 5 | 19.50 (5.29) | 40.83 (10.12)
  Step 6: number analyzed (Participants) | 7 | 5
  Step 6 | 10.0 (13.87) | 36.0 (15.44)
  Step 7: number analyzed (Participants) | 6 | 3
  Step 7 | 4.0 (9.63) | 41.67 (16.41)
  Step 8: number analyzed (Participants) | 4 | 1
  Step 8 | 5.0 (5.0) | 25.0 (NA) — Single data point, no standard error available
  Step 9: number analyzed (Participants) | 1 | 0
  Step 9 | 10.0 (NA) — Single data point, no standard error available |
Statistical Analysis 1: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Goodness of fit test of a two-variable negative binomial multi-level model of maximum distress as a function of step and timepoint. This multi-level model was generated using the menbreg function in Stata 16; Test type: Other — This was a goodness of fit test of a multi-level model, fit was tested using a wald chi-square test; p < .001, Chi-squared — a priori threshold for significance was p=0.05; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; This statistical analysis involved testing of the step-by-timepoint interaction in the two-variable negative binomial model of maximum distress as a function of step and timepoint; Test type: Superiority; p > .05, Mixed Models Analysis — a priori threshold for significance of 0.05
Statistical Analysis 3: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Goodness of fit test of a two-variable negative binomial multi-level model of maximum distress as a function of treatment group and timepoint. This multi-level model was generated using the menbreg function in Stata 16; Test type: Other — This was a goodness of fit test of a multi-level model, fit was tested using a wald chi-square test; p < .001, Chi-squared — a priori threshold for significance of p=0.05; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; This statistical analysis involved testing of the step-by-timepoint interaction in the two-variable negative binomial model of maximum distress as a function of group and timepoint; Test type: Superiority; p < .001, Mixed Models Analysis — a priori threshold for significance of p=0.05
Statistical Analysis 5: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; Goodness of fit test of a two-variable negative binomial multi-level model of maximum distress as a function of step and group. This multi-level model was generated using the menbreg function in Stata 16; Test type: Other — This was a goodness of fit test of a multi-level model, fit was tested using a wald chi-square test; p < 0.001, Chi-squared — a priori threshold for significance was p=0.05; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) vs Control iTBS, Vertex; This statistical analysis involved testing of the step-by-timepoint interaction in the two-variable negative binomial model of maximum distress as a function of step and group; Test type: Superiority; p = 0.024, Mixed Models Analysis — a priori threshold for significance of p=0.05

ADVERSE EVENTS:
Time Frame: Adverse event data were reported over the duration of each subject's participation in the study (i.e. from enrollment to 1 week after the completion of the third TMS treatment).
Description: No difference in definitions. TMS is a low-risk intervention, with the most serious adverse event generally being a seizure (occurring at a rate of approximately 1 in 30,000 in the general population). This study is a low/minimal risk study. Transient stimulation site discomfort was noted in both groups and rated immediately following TMS treatment as seen in outcomes data utilizing the McGill pain questionnaire.
Arm/Group | Active iTBS, Ventromedial Prefrontal Cortex (vmPFC) | Control iTBS, Vertex
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
1. Early termination leading to small numbers of subjects analyzed and limited statistical analysis (in part due to COVID)
2. Equipment limitations and technical problems with physiologic data measurement leading to intermittent unreliable/uninterpretable data
3. Brief duration of treatment contributing to lack of differentiation between experimental groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04019054/Prot_SAP_002.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04019054/ICF_003.pdf